CLINICAL TRIAL: NCT05150860
Title: Communities Fighting COVID!: Returning Our Kids Back to School Safely
Brief Title: Communities Fighting COVID Return to School
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Susan M Kiene, Professor, San Diego State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HS-2021-0208; 1OT2HD108112-01 (NIH)
Record Dates: First submitted 2021-12-03; First posted 2021-12-09 (Actual); Results first posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- At-home testing (Experimental): At-home COVID-19 testing model
  Interventions: Behavioral: At-home COVID-19 testing
- On-site testing (Active Comparator): On-site COVID-19 testing model
  Interventions: Behavioral: Onsite COVID-19 testing

INTERVENTIONS:
Behavioral: At-home COVID-19 testing — At-home over-the-counter (OTC) COVID-19 testing kits provided to middle school students and staff
  Arms: At-home testing
Behavioral: Onsite COVID-19 testing — Onsite COVID-19 testing for middle school students and staff
  Arms: On-site testing

SUMMARY:
San Diego State University (SDSU), a designated Hispanic-serving institution, is partnering with Sweetwater Union High School District, an independent public school district serving 90% ethnic minority and a high proportion of socioeconomically disadvantaged students, and other community partners, to generate evidence for effective and feasible COVID-19 testing for unvaccinated and medically vulnerable middle school students and staff as part of broader COVID mitigation strategies including vaccination to return students back to school safely.

DETAILED DESCRIPTION:
Equitable access to coronavirus 2019 (COVID-19) screening is important to reduce transmission and maintain in-person learning for middle school communities, particularly in disadvantaged schools. Rapid antigen testing, and at-home testing in particular, could offer substantial advantages over onsite testing from a school district's perspective, but it is unknown if engagement in at-home testing can be initiated and sustained. The investigators hypothesized that an at-home COVID-19 school testing program would be non-inferior to an onsite school COVID-19 testing program with regard to school participation rates and adherence to a weekly screening testing schedule. The study enrolled 3 middle schools within a large, predominantly Latinx-serving, independent school district into a noninferiority trial from October 2021 to March 2022. Two schools were randomized to onsite and 1 school to at-home COVID-19 testing programs. All students and staff were eligible to participate.

ELIGIBILITY:
Inclusion Criteria:

* student at a Sweetwater Union High School District Middle School, staff at a Sweetwater Union High School District Middle School

Exclusion Criteria:

* <2 years of age
* Not a student or staff at a participating Sweetwater Union High School District Middle School

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 852 (Actual)
Dates: Start 2021-10-17 (Actual); Primary Completion 2022-04-02 (Actual); Study Completion 2022-04-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Sweetwater Union High School District, Chula Vista, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with the NIH RADx-UP Coordination and Data Collection Center (CDCC). The CDCC is charged by the NIH with making data funded by the RADx-UP initiative available to other researchers. Data are available on the NIH COVID RADx® Data Hub.
Time Frame: Data are available when released by NIH COVID RADx® Data Hub after study completion. Data are available as long as maintained within the Data Hub.
Access Criteria: Researchers can request access to the study data in the Data Hub via dbGaP, where they follow the prompts to request access. Once access is granted, the Researcher will be notified by email. If the Researcher is granted access to a specific study file, they will also have access to all the Data and Metadata files attached to the study.
URL: https://radx-hub.nih.gov/home

REFERENCES:
- [Background] McDaniels-Davidson C, Arechiga-Romero M, Snyder T, Chris N, Sturgis K, Moore V, Bravo R, Famania-Martinez L, Oren E, Kiene SM. Development of an At-Home COVID-19 Test Results-Reporting System for a School District Primarily Serving Underrepresented Minority Groups, San Diego, CA, 2021-2022. Am J Public Health. 2022 Nov;112(S9):S883-S886. doi: 10.2105/AJPH.2022.307073. Epub 2022 Oct 20. PMID 36265090
- [Result] Kiene SM, McDaniels-Davidson C, Lin CD, Rodriguez T, Chris N, Bravo R, Moore V, Snyder T, Arechiga-Romero M, Famania-Martinez L, Carbuccia J, Pinuelas-Morineau R, Oren E. At-Home Versus Onsite COVID-19 School-based Testing: A Randomized Noninferiority Trial. Pediatrics. 2023 Jul 1;152(Suppl 1):e2022060352F. doi: 10.1542/peds.2022-060352F. PMID 37394511
- Available data/document: COVID Rapid Acceleration of Diagnostics (RADx) Data Hub — https://radx-hub.nih.gov/home — Data from this study is available on the RADx Data Hub

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Trial enrollment of participants occurred from mid-October 2021 through late March 2022, with COVID-19 testing occurring from November 7, 2021 to March 27, 2022; the length of possible trial participation varied from 2 to 21 weeks. Participants were recruited from the three participating middle school populations. All students and school staff at the participating schools were eligible to enroll in the trial.
Pre-assignment Details: Schools were excluded if they had a lower proportion of students from households receiving SNAP Program benefits and a lower proportion of underrepresented minority students compared with other schools (3 schools); had ongoing school-wide testing programs with a commercial provider (2 schools); had larger (1 school) or smaller (1 school) student populations (for matching purposes) than the remaining schools; or were geographically closer to the remaining schools (1 school).
Units Other Than Participants: schools
Groups:
- At-home COVID-19 Testing: Weekly COVID-19 screening testing using at-home rapid antigen tests
- Onsite COVID-19 Testing: Weekly COVID-19 screening testing onsite at school with rapid antigen tests
Period: Overall Study
Arm/Group | At-home COVID-19 Testing | Onsite COVID-19 Testing
Started | 264; 1 schools (participants within one school who enrolled in the trial) | 588; 2 schools (participants within 2 schools who enrolled in the trial)
Students | 199; 1 schools | 500; 2 schools
School Staff | 65; 1 schools | 88; 2 schools
Completed | 264; 1 schools | 588; 2 schools
Not Completed | 0; 0 schools | 0; 0 schools

BASELINE CHARACTERISTICS:
Population: Student and school staff participants enrolled in the trial
Groups:
- Total: Total of all reporting groups
Arm/Group | At-home COVID-19 Testing | Onsite COVID-19 Testing | Total
Number analyzed (Participants) | 264 | 588 | 852
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.04 (14.18) | 17.10 (11.55) | 18.01 (12.49)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender Identity: Man | 95 | 251 | 346
  Gender Identity: Woman | 165 | 325 | 490
  Gender Identity: Another category (transgender, genderqueer, bigender, agender) | 4 | 12 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race and ethnicity: Latinx | 218 | 500 | 718
  Race and ethnicity: Filipino, Asian, or Asian Pacific Islander | 9 | 45 | 54
  Race and ethnicity: African American/Black | 3 | 6 | 9
  Race and ethnicity: Another race or ethnicity | 14 | 10 | 24
  Race and ethnicity: Non-Hispanic white | 20 | 27 | 47
Region of Enrollment [Number; unit: participants]
  United States | 264 | 588 | 852
Primary language spoken at home [Count of Participants; unit: Participants]
  Spanish | 66 | 107 | 173
  English | 198 | 481 | 679

OUTCOME MEASURES:

1. Primary Outcome: Adherence to the Weekly COVID-19 Testing Schedule
Description: Proportion of scheduled weekly COVID-19 tests completed when enrolled in the trial
Time Frame: through study completion, up to 21 weeks
Population: Student and school staff participants enrolled in the trial
Measure: Mean (Standard Error); unit: proportion of scheduled tests completed
Arm/Group | At-home COVID-19 Testing | Onsite COVID-19 Testing
Number analyzed (Participants) | 264 | 588
proportion of scheduled tests completed | 0.394 (0.038) | 0.352 (0.032)

ADVERSE EVENTS:
Time Frame: 21 weeks
Arm/Group | At-home COVID-19 Testing | Onsite COVID-19 Testing
All-Cause Mortality (participants affected / at risk) | 0/264 | 0/588
Serious Adverse Events (participants affected / at risk) | 0/264 | 0/588
Other Adverse Events (participants affected / at risk) | 0/264 | 0/588

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-08): https://cdn.clinicaltrials.gov/large-docs/60/NCT05150860/Prot_SAP_000.pdf